CLINICAL TRIAL: NCT00169806
Title: Randall's Plaques: Pathogenesis and Relationship to Nephrolithiasis
Brief Title: Randall's Plaque Study: Pathogenesis and Relationship to Nephrolithiasis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana Kidney Stone Institute (Other)
Collaborators: Indiana University School of Medicine (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, James Lingeman, James Lingeman, MD, Indiana Kidney Stone Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 98-073
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Nephrocalcinosis; Renal Calculi; Hypercalciuria; Hyperparathyroidism; Cystinuria
Keywords: Randall's Plaque; Kidney stones
MeSH Terms: conditions — Nephrocalcinosis; Kidney Calculi; Hypercalciuria; Hyperparathyroidism; Cystinuria | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cohort (Other): Subjects who are scheduled to undergo a percutaneous kidney stone removal who do not have complicated comorbidities
  Interventions: Other: videotape for mapping of renal anatomy and papillary biopsy

INTERVENTIONS:
Other: videotape for mapping of renal anatomy and papillary biopsy — Subjects who enroll in this study will have their renal anatomy videotaped for mapping purposes. Stone location and characteristics will be documented as will papilla and calyces. One or more papillary biopsies will be taken for analysis.

SUMMARY:
Kidney stones are very common. They affect 3-5% of the population in the United States. Many people are hospitalized for the treatment of kidney stones and some may die. Better understanding of what causes kidney stones is useful in both the treatment and prevention of kidney stones. However, exactly what causes kidney stones is unknown.

The most common type of kidney stones contains calcium, which sometimes is attached to a part of the kidney important in producing the final urine, called the papilla. The investigators have noticed that persons who form kidney stones seem to have more papilla with stones attached. They propose to study these areas of the papilla, called Randall's plaques (named after their discoverer), in patients undergoing surgery for kidney stones.

DETAILED DESCRIPTION:
In order to attempt to explain the pathogenesis of renal calculi, the investigators videotape and document the location and characteristics of each stone, papillae and calyces. One or more small papillary biopsies are taken for analysis to help determine the point of origin of the kidney stone and histological studies are undertaken to determine tissue differences amongst different types of stone formers. Approximately one month after surgery, metabolic studies are undertaken to further review potential causes of stone formation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Methodist Urology in Indianapolis, IN who are undergoing endoscopic procedures for nephrolithiasis or other urologic disease.
* Upper urinary tract endoscopic or PERC procedure for kidney stones removal
* General medical health allowing surgical procedure
* Ability to complete all the necessary components of the study
* Able to sign an informed consent

Exclusion Criteria:

* Poor general medical health
* Bleeding diathesis
* Inability or unwillingness to comply with post-surgical follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 1998-11; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To find out why people form stones by comparing 24 urine collections, biopsy and anatomy to other patients who do not form stones and other patients who do form stones to see if the differences are significant | One year from study completion

CONTACTS AND LOCATIONS:
Overall Officials: James Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (1):
- IU Health North Hospital, Indianapolis, Indiana, United States